CLINICAL TRIAL: NCT05675579
Title: A Phase II Study of Neoadjuvant Sacituzumab Govitecan and Pembrolizumab Therapy for Immunochemotherapy-resistant Early-stage Triple-negative Breast Cancer (TNBC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0431; NCI-2022-10926 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — sacituzumab govitecan; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sacituzumab Govitecan and Pembrolizumab (Experimental): Participants will receive drug on Days 1 and 8 of Cycles 1-4, Participants will receive sacituzumab govitecan by vein.
  Participants will receive drug on Days 1, 8, and 15 of each cycle, Participants will receive pembrolizumab by vein.
  Interventions: Drug: Sacituzumab Govitecan; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Sacituzumab Govitecan — Given by IV (vein)
  Other Names: (IMMU-132) Immunomedics
Drug: Pembrolizumab — Given by IV (vein)
  Other Names: KEYTRUDA®

SUMMARY:
To learn if sacituzumab govitecan and pembrolizumab, when given before surgery, can help to control early-stage triple negative breast cancer that has not responded well to other treatments.

DETAILED DESCRIPTION:
Primary Objective:

• To determine the efficacy of sacituzumab govitecan and pembrolizumab combination treatment on pathological complete response (pCR)/residual cancer burden (RCB)-1 in the patients with early-stage TNBC who showed a resistance to the combination of immunochemotherapy.

Secondary Objectives:

* To determine the safety of the proposed combination treatment.
* To determine the objective overall response rate (ORR) of the proposed treatment.
* To determine the distant-recurrence-free survival (DRFS).
* To determine the 3-year event-free survival (EFS) rate.
* To determine the 3-year overall survival (OS) rate.

Exploratory Objective:

• To investigate the response biomarkers in the tumor tissues and peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients 18 years of age or older.
2. Histologically or cytologically confirmed breast cancer
3. T1c N1-2 or T2-4 N0-2 early-stage disease
4. ER/PR negative (ER/PR <1%) or ER/PR low positive (1%≤ER/PR≤10%), and HER2 negative as per institutional and ASCO-CAP guidelines)
5. Initiated the NAC with the first regimen of KN-522 regimen (i.e., pembrolizumab 200 mg Q3W, given with 4 cycles of paclitaxel + carboplatin).
6. ECOG performance score of 0 or 1.
7. The volumetric change of primary tumor = 0% or increase in volumetric size by US or MRI after completing the first part of the KN-522 regimen.
8. Negative serum pregnancy test within 72 hours of receiving the first dose of the study medication for women of childbearing potential as per institutional guidelines. Postmenopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo pregnancy tests.
9. Agreed with undergoing the image-guided core needle biopsy after completing the first part of neoadjuvant treatment regimen.
10. Subjects of childbearing potential should be willing to use effective birth control methods or be surgically sterile or abstain from heterosexual activity for the course of the study through at least 4 months after the last dose of the study drug. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. Effective methods of birth control include:

    * Use hormonal birth control methods: pills, shots/injections, implants (placed under the skin by a health care provider), or patches (placed on the skin).
    * Intrauterine devices (IUDs).
    * Using 2 barrier methods (each partner must use 1 barrier method) with a spermicide. Males must use the male condom (latex or other synthetic material) with spermicide. Females must choose either a Diaphragm with spermicide, cervical cap with spermicide, or a sponge.
11. The patient must have adequate organ function as determined by the following laboratory values:

    * Absolute neutrophil count* ≥ 1,500 /μL
    * Platelets* ≥ 100,000 /μL
    * Hemoglobin* ≥ 9 g/dL
    * Creatinine clearance > 50 ml/min
    * Total bilirubin ≤ 1.5 X ULN
    * Alanine aminotransferase and aspartate aminotransferase < 2.5 X ULN *Hematologic counts above should be without transfusion or growth factor support within 2 weeks of study drug initiation.

Exclusion Criteria:

1. Stage IV disease
2. Any other previous antitumor therapies for the current cancer event.
3. Pregnant or planning to become pregnant during therapy.
4. Gastrointestinal tract disease or defect or previous history of colitis.
5. Has an active autoimmune disease that requires systemic therapy within two years of treatment or a medical condition that requires immunosuppression.
6. Myocardial infarction within 6 months before starting therapy, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication.
7. Has known human immunodeficiency virus (HIV) infection or active hepatitis B or C infection (screen test is not required). Subjects positive for hepatitis C (HCV) antibody are eligible only if the polymerase chain reaction is negative for HCV RNA.
8. Has a cognitive impairment.
9. Any other major comorbidities that can impact receiving immunotherapy or Sacituzumab govitecan.
10. Have live vaccinations within 30 days prior to registration and receive study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Clinton Yam, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org